CLINICAL TRIAL: NCT04143854
Title: Phase II, Randomized, Double-blind, Placebo Controlled, Multi-Center, Dose-ranging and Open Label Extension Clinical Trial to Evaluate the Efficacy and Safety of MBA-P01 in Treatment of Moderate to Severe Lateral Canthal Lines
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of MBA-P01 in Treatment of Lateral Canthal Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT14-AU18LCL209
Record Dates: First submitted 2019-10-28; First posted 2019-10-29 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Lateral Canthal Lines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBA-P01 24U (Experimental): Experimental group; Dose: 24U
  Interventions: Drug: MBA-P01(Botulinum toxin A)
- MBA-P01 12U (Experimental): Experimental group; Dose: 12U
  Interventions: Drug: MBA-P01(Botulinum toxin A)
- Placebo (Placebo Comparator): Placebo group; normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MBA-P01(Botulinum toxin A) — Intramuscular injection; Dose varies by group
  Arms: MBA-P01 12U; MBA-P01 24U
Drug: Placebo — Intramuscular injection; normal saline
  Arms: Placebo

SUMMARY:
This phase 2 study includes two treatment period; 1)Dose- ranging period, Day 0 to 16 weeks, which will assess dose-related safety/tolerance, and the potential to improve the appearance of lateral canthal lines and 2) open-label extension period, 16 weeks to 52 weeks, which will evaluate the long term-safety of MBA-P01

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65
* Bilaterally symmetrical moderate to severe lateral canthal lines(LCLs) at maximum smile as assessed by both investigator and subject using FWS

Exclusion Criteria:

* History of facial nerve paralysis
* Any eyebrow or eyelied ptosis as determined by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Facial wrinkle scale(FWS) change of lateral canthal line at maximum smile | 4 weeks
  Proportion of subjects achieving at least a 2 grade decrease from baseline and a grade 0 or 1 in Facial Wrinkle Scale (0: none to 3: severe) of LCL at maximum smile, as assessed by the investigator and subject

CONTACTS AND LOCATIONS:
Locations (1):
- Maroubra Medical Centre, Maroubra, New South Wales, Australia